CLINICAL TRIAL: NCT00481208
Title: Diurnal Intraocular Pressure and Peripapillary Retinal Blood Flow in Medically Controlled Open-Angle Glaucoma
Acronym: IOPMG
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Other Study IDs: 4-2006-0146
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Open-Angle Glaucoma
Keywords: open-angle glaucoma; diurnal fluctuation; intraocular pressure; peripapillary retinal blood flow; latent asymmetric intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Diurnal fluctuations of intraocular pressure (IOP) and peripapillary retinal blood flow may have distinctive patterns in medically well-controlled open-angle glaucoma patients. In the results, we found a unique pattern, 'Latent asymmetric IOP', defined as the IOP which differs between the eyes only when placed in the supine position. Unique effects of this latent asymmetric IOP on Visual field and diurnal IOP fluctuations were studied.

DETAILED DESCRIPTION:
Diurnal fluctuations of intraocular pressure (IOP) and peripapillary retinal blood flow have been implicated to be one of the important factors to affect visual field progression. However, there was no study to investigate them in medically well-controlled open-angle glaucoma patients. So we want to find the unique patterns.

Study 1. Subjects : Patients with medically well controlled open angle glaucoma Method : IOP and peripapillary retinal blood flow were measured for 24 hours. The relationship between the two were studied.

Study 2. Of the patients enrolled in study 1 , those on the same medical regimen for both eyes were analyzed for the presence of a latent asymmetric IOP and it's influence and association with visual field and diurnal IOP fluctuation.

ELIGIBILITY:
Inclusion Criteria:

* Open-angle glaucoma
* Topical anti-glaucoma medications

Exclusion Criteria:

* Ocular surgery history
* Other ocular disease history
* Oral glaucoma medications

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-03; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chan Yun Kim, MD, PhD, Study Chair — Department of Ophthalmology, Yonsei University College of Medicine
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea